CLINICAL TRIAL: NCT02765737
Title: Dehydrated Human Amnion Chorion Membrane (dHACM) vs. Control in the Treatment of Partial Thickness Burns.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment, issues with inclusion/exclusion and choice of control
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFBUR002
Record Dates: First submitted 2016-05-05; First posted 2016-05-09 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2020-11

CONDITIONS: Treatment of Partial Thickness Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Treatment 1 - dHACM plus Control Burn Area A Treatment 2 - Control Burn Area B
  Interventions: Other: Dehydrated Human Amnion/Chorion Membrane; Device: Mepilex Ag
- Group 2 (Active Comparator): Treatment 1 - dHACM plus Control Burn Area B Treatment 2 - Control Burn Area A
  Interventions: Other: Dehydrated Human Amnion/Chorion Membrane; Device: Mepilex Ag

INTERVENTIONS:
Other: Dehydrated Human Amnion/Chorion Membrane — Dehydrated human amnion/chorion membrane (dHACM) product and is regulated as a Human Cells, Tissues and Cellular and Tissue Based Product (HCT/P) under Section 361 of the Public Health Service Act by the Food and Drug Administration (FDA).
  Other Names: dHACM
Device: Mepilex Ag

SUMMARY:
Multicenter, prospective, randomized, controlled feasibility trial to determine the safety and effectiveness of Dehydrated Human Amnion Chorion Membrane (dHACM) plus Control as compared to Control alone for the treatment of second degree burns (partial thickness burns) as assessed by time to healing and scarring

DETAILED DESCRIPTION:
Multicenter, prospective, randomized, controlled feasibility trial to determine the safety and effectiveness of Dehydrated Human Amnion Chorion Membrane (dHACM) plus Control as compared to Control alone for the treatment of second degree burns as assessed by time to healing and scarring

ELIGIBILITY:
Inclusion Criteria:

ll patients enrolled must meet all the following criteria:

1. Patient with burn injury that meets all of the following requirements:

   1. Occurred within the last 48 hours
   2. Wound is thermal in nature
   3. Partial-thickness burn (burn extends through the epidermis and may penetrate into the dermis)
   4. Total body surface area (TBSA) of burn(s) is 2-20% for all subjects
   5. Burn area(s) located on smooth, flat surface
   6. 2 burn areas, each with a minimum size of 16cm2 (burn areas may be two separate burns or within one large burn, see Section 9.4.2)
2. Age ≥ 12 months and ≤ 70 years

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded:

1. Burns meeting any of the following criteria:

   1. Mechanism of injury was electrical, radiation, chemical or frostbite
   2. Wound is larger than 200 cm2
   3. Clinically infected burn (as judged by the investigator)
   4. Previous or planned treatment of the Burn Area(s) with any of the following:

      * Biological Skin Substitutes (including Apligraf®, Dermagraft®, etc.)
2. Patient criteria that will make patient ineligible for enrollment:

   1. Ventilator dependence
   2. Active malignant disease or patient is less than 1 year disease-free
   3. Use of immunosuppressive agents, radiation or chemotherapy within the past 30 days
   4. Auto-immune disorders including Systemic Lupus Erythematosus (SLE), Fibromyalgia, Acquired Immunodeficiency Syndrome (AIDS) or Human Immunodeficiency Virus (HIV)
   5. Presence of any condition (including current drug or alcohol abuse, medical or psychiatric condition) that is likely to impair understanding of or compliance with the study protocol in the judgment of the Investigator
   6. Presence of any condition that is likely to compromise healing in the judgment of the Investigator
   7. Pregnancy at enrollment or within last 6 months, women who are breastfeeding, or women of childbearing potential who are planning to become pregnant during the time of the study OR are unwilling/unable to use acceptable methods of contraception (birth control pills, barriers, or abstinence)
   8. Patient has been on any investigational drug(s) or therapeutic device(s) in the last 30 days or any previous enrollment in this study
3. Allergy or known sensitivity to any of the following:

   1. Aminoglycosides such as gentamicin sulfate and/or streptomycin sulfate
   2. Silver

      -

Ages: 12 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-04; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Healing Rate | 3 weeks
  95% epitheliazation as assesses by the investigator
Freedom from Scarring | 3 Months
  Vancouver Scar Scale: consists of four variables: pliability, vascularity, height (thickness), and pigmentation. Each variable has four to six possible scores. A total score ranges from 0 to 14, whereby a score of 0 reflects normal skin.

SECONDARY OUTCOMES:
Reduction in pain | 3 weeks
  Visual Analog Scale or FLACC Behavioral Pain Assessment Scale:VAS-No pain on left of line, worst pain imaginable on the right of line; FLACC- 0-2, (0 being least uncomfortable to 2 which is very uncomfortable)

CONTACTS AND LOCATIONS:
Overall Officials: David Mason, MD, Study Director — Chief Medical Officer
Locations (6):
- United States (6):
  - Arizona Burn Center, Phoenix, Arizona
  - Keck School of Medicine, Los Angeles, California
  - University of San Diego Nedical Center, San Diego, California
  - St Elizabeth Reg Med Center, Lincoln, Nebraska
  - Bruce Cairns Surgery Burn Center, Chapel Hill, North Carolina
  - Drexel University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No